CLINICAL TRIAL: NCT03383068
Title: Research of Intensive Metabolic Intervention Before Pregnancy in Polycystic Ovary Syndrome
Brief Title: Research of Intensive Metabolic Intervention Before Pregnancy in PCOS
Acronym: PCOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2017]055
Record Dates: First submitted 2017-11-28; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: PCOS; Impaired Glucose Tolerance
Keywords: PCOS; imparied glucose tolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Acarbose; Exenatide; Orlistat; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- control (Other): metformin(1000-1500mg/d) treated for 6 months, reverse to normal glucose tolerance
  Interventions: Drug: Metformin
- acarbose (Experimental): metformin(1000-1500mg/d) treated for 6 months, can not reverse to normal glucose tolerance, then treat with acarbose (100mg tid ) for 3 months
  Interventions: Drug: Acarbose 100 MG
- Exenatide (Experimental): metformin(1000-1500mg/d) treated for 6 months, can not reverse to normal glucose tolerance, then treat with Exenatide 10μg/bid ) for 3 months
  Interventions: Drug: Exenatide
- Orlistat (Experimental): metformin(1000-1500mg/d) treated for 6 months, can not reverse to normal glucose tolerance, then treat with Orlistat(0.12mg/tid ) for 3 months
  Interventions: Drug: Orlistat

INTERVENTIONS:
Drug: Acarbose 100 MG — for metformin uneffective subjects, using acarbose for 3 months
  Other Names: Acarbose
  Arms: acarbose
Drug: Exenatide — for metformin uneffective subjects, using Exenatide for 3 months
  Arms: Exenatide
Drug: Orlistat — for metformin uneffective subjects, using Orlistatfor 3 months
  Arms: Orlistat
Drug: Metformin — metformin effective subjects,act as control group
  Other Names: METF
  Arms: control

SUMMARY:
To investigate whether intensive metabolic intervention of PCOS women before pregnancy can improve pregnancy outcome.Besides, the investigators aim to investigate the best therapy strategy of metabolic intervention before pregnancy.The investigators plan to recruit PCOS women at childbearing age. By using acarbose, GLP-1 analogue, berberin et al. the investigators will intervent the participants' metabolic statues for 3 months before pregnancy and to compare outcome in each group.

DETAILED DESCRIPTION:
To investigate whether intensive metabolic intervention of PCOS women before pregnancy can improve pregnancy outcome.Besides, the investigators aim to investigate the best therapy strategy of metabolic intervention before pregnancy.The investigators plan to recruit PCOS women with IGR / DM not effective of metformin treatment at childbearing age. By using acarbose, GLP-1 analogue, berberin et al. the investigators will intervent the participants' metabolic statues for 3 months before pregnancy and to compare outcome in each group.

ELIGIBILITY:
Inclusion Criteria:

* PCOS women at Childbearing Age
* PCOS: Clinical hyperandrogenism and/or hyperandrogenemia, menstrual dysfunction (oligomenorrhea or amenorrhea) and exclusion of other known disorders. PCOS will be diagnosed using the 2003 Rotterdam criteria.

Exclusion Criteria:

* Past or present history of a medical disorder or medication known to affect body composition, insulin secretion and sensitivity, or the growth hormone (GH)-insulin-like growth factor 1 (IGF1) axis (eg steroid hormone or thyroid replacement).
* History of current or past pregnancy
* Hormonal contraceptive or metformin use within 3 months of enrollment
* Nonclassical congenital adrenal hyperplasia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of pregnant rate after intensive metabolic intervention | up to 24 weeks
  To compare the pregnant rate of four groups after treatment

SECONDARY OUTCOMES:
Improvement of obsorbtion rate after intensive metabolic intervention | up to 24 weeks
  To compare the obsorbtion rate of four groups after treatment
Improvement of stillborn foetus rate after intensive metabolic intervention | up to 24 weeks
  To compare the stillborn foetus rate of four groups after treatment
Improvement of hyperandrogenism | up to 24 weeks
  To compare the free androgen index of three groups after treatment
Improvement of intravenous blood glucose from impaired glucose regulation to normal glucose regulation | up to 24 weeks
  To compare the intravenous blood glucose of three groups after treatment
Improvement of triglyceride | up to 24 weeks
  To compare the circulating triglyceride of three groups after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Department of Endocrinology and Metabolism, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No